CLINICAL TRIAL: NCT04861116
Title: AcAdeMiC: Acting With Acceptance, Mindfulness and Compassion to Overcome Test/Exam Anxiety - An ICT-based Psychotherapeutic Intervention for Adolescents
Brief Title: AcAdeMiC: Acting With Acceptance, Mindfulness and Compassion to Overcome Test/Exam Anxiety
Acronym: AcAdeMiC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Cláudia Pires, Principal Investigator, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFRH/BD/143520/2019
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Adolescents; Test Anxiety
Keywords: test anxiety; adolescents; acceptance; mindfulness; compassion
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention program for test anxiety (Experimental): 12 weekly ICT-delivered individual sessions.
  Interventions: Behavioral: Intervention program for test anxiety
- Control (No Intervention): Waiting list that will have access to the intervention program after the 6-month follow-up assessment.

INTERVENTIONS:
Behavioral: Intervention program for test anxiety — 12-week ICT-based manualized, targeted and facilitated individual intervention for adolescent students, that aims to promote compassion, acceptance and mindfulness, in order to help improve test anxiety's regulation (and consequently symptom reduction), as well as increase general and school-related well-being, while promoting valued life action.
  Other Names: AcAdeMiC: Acting With Acceptance, Mindfulness and Compassion to Overcome Test/Exam Anxiety
  Arms: Intervention program for test anxiety

SUMMARY:
Test Anxiety is a highly prevalent and impairing condition in adolescents (i.e., 9th to 12th grade students), significantly impacting on their mental health and well-being. Among Portuguese university students, test anxiety is the primary reason for seeking specialized psychological support, suggesting the importance of early intervention.

Test anxiety associates to low self-compassion, acceptance and mindfulness, which have been increasingly acknowledged in literature as important processes to cultivate towards human experience and suffering, within intervention programs, particularly in adolescence, and in anxiety and fear of failure in academic settings.

These processes are covered and enhanced within comprehensive models and evidence-based therapies that adopt an integrative, contextual and biopsychosocial approach, such as Acceptance and Commitment Therapy (ACT), and Mindfulness-Based Cognitive Therapy (MBCT), as well as an evolutionary approach, such as Compassion Focused Therapy (CFT). These approaches focus on receiving internal events (e.g., thoughts, emotions, memories) in an accepting and compassionate way, as part of human experience, without changing them, while developing a sense of vitality, well-being and commitment to valued ends in life, instead of focusing solely or mainly on symptom reduction (although it is usually a consequent outcome).

However, there are no empirically validated therapeutic programs for adolescents with test anxiety promoting these processes combined.

ICT-based interventions are accessible, convenient, cost-effective and have been proved effective in reducing anxiety disorders' symptomatology. Even though there are some empirically validated online interventions for test anxiety in adolescents, having shown promising results, these were mainly self-help/module-based programs, without a clinician facilitating the intervention.

This project aims to develop and implement a 12-week ICT-based targeted, facilitated and manualized individual intervention for adolescent students, developing compassion, acceptance and mindfulness, in order to help improve test anxiety's regulation (and consequently symptom reduction), as well as increase general and school-related well-being, while promoting valued life action.

DETAILED DESCRIPTION:
All ethical and deontological requirements are guarenteed in this study.

A sample of adolescent students (from 9th to 12th grade) is being online-recruited, through social media and contacts with Executive Boards of Portuguese secondary schools, private practices and study centers, advertising the study.

Parents/legal guardians are encouraged to contact the team. From this approach, parents/legal guardians and respective adolescents who demonstrate interest are explained the aims and procedures of the study and asked to sign a written consent form.

Adolescents are then assessed for eligibility through a test anxiety self-report measure and a clinical interview.

Eligible participants will be randomly assigned to either an experimental group, who will reveive the intervention (facilitated by licenced psychotherapists with training in contextual therapies and are familiar with the intervention protocol), or a waiting-list control group, who will have access to the intervention after the six-month follow-up assessment.

Both groups will complete a protocol with self-report measures, assessing psychopathology indicators, emotion regulation processes, and general and school-related well-being, in four different moments: at baseline (M0), immediatly after the intervention (M1), three months (M2) and six months (M3) after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* provision of written informed consent by participants and their legal guardians;
* presence of high levels of test anxiety, confirmed through self-report assessment and clinical interview;
* educational level from 9th to 12th grade;
* absence of Neurodevelopmental Disorders, except Specific Learning Disorders of mild severity;
* absence of any degree of cognitive decline or impairment;
* absence of any severe Depressive Disorder;
* absence of any other severe psychiatric condition (e.g., Obsessive-Compulsive Disorder, Bipolar Disorder, Psychotic Disorders);
* not being under treatment for a psychiatric condition.

Exclusion Criteria:

* no provision of written informed consent by participants and their legal guardians;
* absence of high levels of test anxiety, confirmed through self-report assessment;
* educational level below 9th and above 12th grade;
* presence of Neurodevelopmental Disorders, except Specific Learning Disorders of mild severity;
* presence of any degree of cognitive decline or impairment;
* presence of any severe Depressive Disorder;
* presence of any other severe psychiatric condition (e.g., Obsessive-Compulsive Disorder, Bipolar Disorder, Psychotic Disorders);
* being under treatment for a psychiatric condition.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Test Anxiety | 6 months [From Baseline to 6 months follow-up]
  Reactions to Tests for Adolescents (RT-A). Participants rate the items on a Likert scale from 1 to 4. Lower scores indicate a better outcome

SECONDARY OUTCOMES:
General well-being | 6 months [From Baseline to 6 months follow-up]
  Mental Health Continuum - Short Form - for Youth (MHC-SF). Participants rate the items on a Likert scale from 0 to 5. Higher scores indicate a better outcome
School-related well-being | 6 months [From Baseline to 6 months follow-up]
  School-related Well-Being Scale (SWBS). Participants rate the items on a Likert scale from 1 to 5. Higher scores indicate a better outcome
Psychological flexibility in test situations | 6 months [From Baseline to 6 months follow-up]
  Test Anxiety Acceptance and Action Questionnaire for Adolescents (TA-AAQ-A). Participants rate the items on a Likert scale from 1 to 7. Higher scores indicate a better outcome
General psychological flexibility | 6 months [From Baseline to 6 months follow-up]
  Avoidance and Fusion Questionnaire for Youth (AFQ-Y). Participants rate the items on a Likert scale from 0 to 4. Lower scores indicate a better outcome
Mindfulness | 6 months [From Baseline to 6 months follow-up]
  Child and Adolescent Mindfulness Measure (CAMM). Participants rate the items on a Likert scale from 0 to 4. Higher scores indicate a better outcome
Self-compassion | 6 months [From Baseline to 6 months follow-up]
  Self-Compassion Scale (SCS-A). Participants rate the items on a Likert scale from 1 to 5. Higher scores indicate a better outcome

OTHER OUTCOMES:
Depression, anxiety and stress | 6 months [From Baseline to 6 months follow-up]
  Depression Anxiety and Stress Scales (DASS-21). Participants rate the items on a Likert scale from 0 to 3. Lower scores indicate a better outcome
Self-criticism | 6 months [From Baseline to 6 months follow-up]
  Forms of Self-Criticizing/attacking and self-Reassuring Scale (FSCRS-A). Participants rate the items on a Likert scale from 0 to 4. Lower scores indicate a better outcome
Shame | 6 months [From Baseline to 6 months follow-up]
  External and Internal Shame Scale for adolescents (EISS-A). Participants rate the items on a Likert scale from 0 to 4. Lower scores indicate a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Cláudia P. Pires, M.Sc., Principal Investigator — University of Coimbra
Locations (1):
- University of Coimbra, Coimbra, Portugal